CLINICAL TRIAL: NCT02567916
Title: A Comparison of Injection Pain of Propofol During Endoscopy : LCT Propofol vs MCT/LCT Propofol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Soo Kim, MD, PhD, Associate Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-08-026-001
Record Dates: First submitted 2015-03-23; First posted 2015-10-05 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Pain; Complication of Injection
MeSH Terms: conditions — Pain | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- FRESOFOL MCT (Experimental): To compare the incidence and intensity of pain on injection that is caused by propofol (LCT propofol) versus fresofol (MCT/LCT propofol) .
  Interventions: Drug: Fresofol
- Propofol (Active Comparator): The purpose of this study is to compare the incidence and intensity of possible pain on injection as well as patient satisfaction caused by propofol (LCT propofol) versus fresofol (MCT/LCT propofol).
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Fresofol
  Arms: FRESOFOL MCT
Drug: Propofol
  Arms: Propofol

SUMMARY:
The purpose of this study is to compare the incidence and intensity of possible pain on injection as well as patient satisfaction caused by long chain triglyceride propofol versus medium/long chain combinated triglyceride propofol on endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* age >15 yrs
* ASA (American Society of Anesthesiologists risk class III-IV)I-II
* patients undergoing to gastroscopy

Exclusion Criteria:

* significant systemic disease (American Society of Anesthesiologists risk class III-IV)
* history of allergic reactions to any of the study drugs
* chronic use of opioid analgesics
* psychiatric disorder
* arrythmia
* pregnancy
* age <18 yrs

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Incidence and Intensity of Pain on Injection That is Caused by Propofol (LCT propofol) Versus the Fresofol (MCT/LCT propofol). | 2 hours

SECONDARY OUTCOMES:
Patient Satisfaction With Sedation Including the Recall of Pain. | 2 hours and 5-7days after the end of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Eun Soo Kim, MD, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- Keimyung University Dongsan Medical Center, Daegu, South Korea

REFERENCES:
- [Background] Ozawa A, Isono M, Ueno T, Kosaka Y, Nakano T, Inamura M, Kanai A, Okamoto H, Hoka S, Nomiyama S. [Comparison of propofol LCT and propofol MCT/LCT regarding the injection pain at different sites and the memory]. Masui. 2005 Nov;54(11):1241-6. Japanese. PMID 16296361